CLINICAL TRIAL: NCT04604132
Title: A Phase 1b/2 Study of Derazantinib as Monotherapy and Combination Therapy With Paclitaxel, Ramucirumab or Atezolizumab in Patients With HER2-negative Gastric Adenocarcinoma Expressing FGFR2 Genetic Aberrations
Brief Title: Derazantinib Alone or in Combination With Paclitaxel, Ramucirumab or Atezolizumab in Gastric Adenocarcinoma
Acronym: FIDES-03
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated prematurely for administrative reasons not related to patient safety.
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZB-CS-202
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Gastric Adenocarcinoma
Keywords: gastric cancer; gastro-esophageal adenocarcinoma; adenocarcinoma of the stomach or gastro-esophageal junction; fibroblast growth factor receptor; FGFR genetic aberration; targeted therapy; derazantinib; atezolizumab; Tecentriq; paclitaxel; ramucirumab; Cyramza; solid tumor
MeSH Terms: conditions — Stomach Neoplasms; Acrocephalosyndactylia | interventions — derazantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Substudy 1: Cohort 1.1 Derazantinib 300 mg once daily (Experimental): Patients with FGFR2 fusions or amplifications were treated with 300 mg Derazantinib monotherapy once daily
  Interventions: Drug: Derazantinib
- Substudy 1: Cohort 1.2 Derazantinib 300 mg once daily (Experimental): Patients with FGFR1-3 mutations were treated with 300 mg Derazantinib monotherapy once daily
  Interventions: Drug: Derazantinib
- Substudy 1: Cohort 1.3 Derazantinib 200 mg twice daily (Experimental): Patients with FGFR fusions, amplifications or mutations were treated with 200 mg Derazantinib monotherapy twice daily
  Interventions: Drug: Derazantinib
- Substudy 2: Derazantinib 200 mg once daily +Paclitaxel+ Ramucirumab (Experimental): Patients with FGFR fusions, amplifications or mutations were treated with 200 mg Derazantinib once daily in combination with Paclitaxel and Ramucirumab
  Interventions: Drug: Derazantinib-paclitaxel-ramucirumab combination
- Substudy 2: Derazantinib 300 mg once daily+Paclitaxel+ Ramucirumab (Experimental): Patients with FGFR fusions, amplifications or mutations were treated with 300 mg Derazantinib once daily combination with Paclitaxel and Ramucirumab
  Interventions: Drug: Derazantinib-paclitaxel-ramucirumab combination

INTERVENTIONS:
Drug: Derazantinib — Derazantinib was administered orally at a dose of 300 mg once daily as monotherapy in the Substudy 1 (Cohort 1.1).
  Arms: Substudy 1: Cohort 1.1 Derazantinib 300 mg once daily
Drug: Derazantinib-paclitaxel-ramucirumab combination — Derazantinib was administered orally at a dose of 200 mg once daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
  Arms: Substudy 2: Derazantinib 200 mg once daily +Paclitaxel+ Ramucirumab
Drug: Derazantinib-paclitaxel-ramucirumab combination — Derazantinib was administered orally at a dose of 300 mg once daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
  Arms: Substudy 2: Derazantinib 300 mg once daily+Paclitaxel+ Ramucirumab
Drug: Derazantinib — Derazantinib was administered orally at a dose of 200 mg twice daily as monotherapy in the Substudy 1 (Cohort 1.3).
  Arms: Substudy 1: Cohort 1.3 Derazantinib 200 mg twice daily
Drug: Derazantinib — Derazantinib was administered orally at a dose of 300 mg once daily as monotherapy in the Substudy 1 (Cohort 1.2).
  Arms: Substudy 1: Cohort 1.2 Derazantinib 300 mg once daily

SUMMARY:
The purpose of this study was to evaluate the efficacy of derazantinib monotherapy or derazantinib in combination with paclitaxel and ramucirumab in patients with gastric adenocarcinoma (GAC) i.e. with human epidermal growth factor receptor 2 (HER2)-negative adenocarcinoma of the stomach or gastro-esophageal junction harboring fibroblast growth factor receptor 2 (FGFR2) genetic aberrations (GA).

DETAILED DESCRIPTION:
The study comprised two open-label substudies in patients with HER2-negative adenocarcinoma of the stomach or gastro-esophageal junction harboring FGFR2 gene translocations, FGFR2 gene amplifications, or FGFR1-3 mutations.

In Substudy 1, GAC patients with specified FGFR GAs, after either first- or second-line treatment, and no approved treatment alternative were treated with derazantinib 300 mg once daily or 200 mg twice daily, with the aim of evaluating the safety, tolerability, and efficacy of derazantinib monotherapy in this patient population.

In Substudy 2, GAC patients with specified FGFR GAs after standard first-line treatment, were treated with a derazantinib-paclitaxel-ramucirumab combination with the aim of evaluating the safety, tolerability, and efficacy of the combination therapy and determining the recommended phase 2 dose (RP2D).

The study originally planned to include three substudies but was prematurely terminated for administrative reasons before the third substudy (including combination therapy with derazantinib plus atezolizumab) was initiated.

ELIGIBILITY:
Main inclusion criteria

Patients meeting all of the inclusion criteria at screening were eligible for enrollment in the study, including:

1. Histologically-confirmed adenocarcinoma of the gastro-esophageal junction or stomach.
2. Negative HER2 status obtained from the most recent available tissue sample.
3. Inoperable recurrent, locally advanced adenocarcinoma or progressing stage IV adenocarcinoma of the gastro-esophageal junction or stomach, and prior anti-tumor treatment as specified for each Substudy. Patients were required to be staged as inoperable at the time of screening in order to avoid interference of any potentially planned surgery with RECIST requirements during the study:

   Substudy 1: Patients with radiographically documented disease progression after either standard first- or second-line treatment, and no approved and/or tolerable treatment alternative.

   Substudy 2: Patients with radiographically documented disease progression after standard first-line treatment, and per Investigator assessment considered suitable to tolerate the treatment regimen.
4. Eligible FGFRfus/amp/mt positive test result. For Substudy 1 Cohort 1.1, FGFR2fus/amp; for Cohort 1.2, FGFR1-3mt; for Cohort 1.3, FGFRfus/amp/mt. For Substudy 2, FGFRfus/amp/mt.
5. Measurable disease as defined by the Investigator using RECIST 1.1 criteria
6. Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1
7. Adequate organ functions as indicated by Screening visit laboratory values.

Main exclusion criteria

Patients meeting any of the following exclusion criteria at screening were not eligible to be enrolled in the study:

* Receipt of prior cancer treatment within specific interval periods.
* For patients enrolled in Substudy 1, prior treatment with FGFR inhibitors.
* For patients enrolled in Substudy 2, prior treatment with:

  * Taxanes within 6 months prior to randomization
  * FGFR inhibitors or pathway-targeting agents
  * Anti-VEGF(R) therapeutic antibody or pathway-targeting agents
* Concurrent evidence of clinically significant corneal or retinal disorder likely to increase the risk of eye toxicity, including but not limited to bullous/band keratopathy, keratoconjunctivitis (unless keratoconjunctivitis sicca), corneal abrasion (unless related to trauma), inflammation/ulceration, confirmed by ophthalmological examination.
* History of clinically significant cardiac disorders, including myocardial infarction, or New York Heart Association Class II to IV congestive heart failure, within 6 months of the first dose of study drug, and/or any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months of the first dose of study drug, and/or concurrent and clinically significant abnormalities on ECG at Screening, including QTcF > 450 ms for males or > 460 ms for females (mean values from triplicate ECGs).
* Any unresolved (at the time of Screening) clinically significant CTCAE Grade ≥ 2 toxicity (except for alopecia, Grade ≤ 2 platinum-therapy related neuropathy, or Grade ≤ 2 anemia from previous anti-tumor treatment and/or from medical/surgical procedures/interventions).
* Known central nervous system metastases.
* Severe bacterial, fungal, viral and/or parasitic infections on therapeutic oral or IV medication at the time of first dose of study drug administration.
* Significant gastrointestinal disorders that could interfere with the absorption, metabolism, or excretion of derazantinib.
* History of additional malignancy that was progressing or required active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Häckl, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (81):
- United States (2):
  - AdventHealth Cancer Institute, Orlando, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Argentina (2):
  - Fundación Favaloro para la Docencia e Investigación Médica, Buenos Aires
  - Hospital de Gastroenterologia Dr. Carlos Bonorino Udaondo, Ciudad Autonoma Buenos Aires
- Australia (3):
  - Monash Medical Centre Clayton, Clayton
  - Peter MacCallum Cancer Centre, Melbourne
  - The Alfred Hospital, Prahran
- Belgium (3):
  - UZA, Edegem
  - UZ Leuven, Leuven
  - AZ Delta, Menen
- Brazil (5):
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal, Rio Grande do Norte
  - Fundação Doutor Amaral Carvalho, Jaú
  - Instituto Nacional de Câncer José Alencar Gomes da Silva, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
- Chile (3):
  - CeCim Biocinetic, Santiago, Region Met
  - Centro de Estudios Clínicos SAGA, Santiago
  - Instituto Clinico Oncologico, Temuco
- France (6):
  - Institut Sainte Catherine, Avignon
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Centre Georges François Leclerc, Dijon
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Staedtisches Klinikum Dresden Standort Dresden-Friedrichstadt, Dresden
  - Krankenhaus Nordwest GmbH, Frankfurt
  - Uniklinik Mainz, Mainz
- Italy (8):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Istituto Clinico Humanitas, Rozzano
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Poland (4):
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - Examen sp. z o.o., Skórzewo
  - Centrum Zdrowia MDM, Warsaw
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Russia (9):
  - SAIH "Republican Clinical Oncological Dispensary of the Ministry of Healthcare of Republic Tatarstan, Kazan'
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - "VitaMed" LLC, Moscow
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - FSBI "Clinical Research and Practical Center for specialized medical care (oncology)", Pesochnyy
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
  - Tomsk Research Instutite of Oncology, Tomsk
  - SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa
- South Korea (8):
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (8):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Turkey (Türkiye) (8):
  - Baskent University Adana Application and Research Center, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet Uni Goztepe Training&Res Hosp, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
- United Kingdom (6):
  - Addenbrooke's Hospital, Cambridge
  - Ninewells Hospital, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London Hospitals, London
  - The Christie, Manchester
  - Royal Marsden Hospital- Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 6 Oct. 2020 to 10 Jun. 2022, 919 patients (pt.) had molecular pre-screening. 66 had clinical screening, and 47 were treated.
  In Substudy 2, pt. were allocated to 1 of 3 dose levels using a dose escalation scheme: Derazantinib at a dose of 200 mg once daily, 300 mg once daily, or 200 mg twice daily, all in combination with paclitaxel and ramucirumab. However, no pt. received the highest dose, therefore only the 200 and 300 mg once daily dose levels are presented in the results section.
Groups:
- Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily; Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily: Derazantinib was administered orally at a dose of 300 mg once daily as monotherapy in the Substudy 1.
- Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily: Derazantinib was administered orally at a dose of 200 mg twice daily as monotherapy in the Substudy 1.
- Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of 200 mg in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
- Substudy 2: Derazantinib 300 mg Once Daily + Paclitaxel + Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of 300 mg in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Period: Overall Study
Arm/Group | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily + Paclitaxel + Ramucirumab
Started | 13 | 8 | 13 | 6 | 7
Completed (One patient still received derazantinib while the study was early terminated and was transferred to a post-trial access program.) | 0 | 0 | 0 | 0 | 1
Not Completed | 13 | 8 | 13 | 6 | 6
Not completed — Adverse Event | 2 | 0 | 0 | 1 | 2
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease: Clinical progression | 0 | 0 | 1 | 0 | 0
Not completed — Progressive disease: Radiological progression | 8 | 7 | 10 | 4 | 3
Not completed — Death | 3 | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily+Paclitaxel+ Ramucirumab | Total
Number analyzed (Participants) | 13 | 8 | 13 | 6 | 7 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.77) | 66.1 (9.39) | 54.8 (13.43) | 55.2 (10.53) | 52.0 (11.34) | 59.3 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 1 | 1 | 5 | 14
  Male | 8 | 6 | 12 | 5 | 2 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 2 | 0 | 2 | 9
  Black/African American | 0 | 0 | 1 | 0 | 0 | 1
  White | 9 | 7 | 9 | 6 | 5 | 36
  Missing | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Substudy 1 (in Cohorts 1.1 and 1.2)
Description: ORR was defined by the percentage of patients with confirmed complete response (CR, which means disappearance of all target lesions) or partial response (PR, which means >=30% decrease in the sum of the longest diameter of target lesions) by blinded independent central review (BICR) using the internationally recognized criteria for the radiological assessment in tumor response of solid tumors (RECIST 1.1). Overall Response (OR) = CR + PR.
  The patients in Cohort 1.1 had FGFR2 fusions or amplification gastric adenocarcinoma (GAC) and FGFR1-3 mutations GAC in Cohort 1.2.
Time Frame: From first dose and up to 18 months
Population: Modified intent-to-treat (mITT) population: all patients who received at least one dose of derazantinib and had at least one post-baseline imaging assessment in accordance with RECIST 1.1 or documented clinical progression or died from any cause on or after the first dose of study treatment and until safety follow-up visit (inclusive).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily
Number analyzed (Participants) | 13 | 8
Percentage of participants | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 31.2]

2. Primary Outcome: Progression-free Survival at 4 Months (PFS4) in Substudy 1 in Cohort 1.3
Description: PFS4 was defined by the percentage of patients alive and free of disease progression (defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions) by BICR per RECIST. 1.1. Patients in this Cohort had FGFR fusions, amplifications or mutations GAC
Time Frame: From first dose and up to 4 months
Population: mITT population: all patients who received at least one dose of derazantinib and had at least one post-baseline imaging assessment in accordance with RECIST 1.1 or documented clinical progression or died from any cause on or after the first dose of study treatment and until safety follow-up visit (inclusive).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 13
Percentage of participants | 7.7 [0.4 to 31.6]

3. Primary Outcome: Recommended Phase 2 Dose (RP2D) in Substudy 2 (Derazantinib-paclitaxel-ramucirumab in Combination)
Description: RP2D was determined from safety and tolerability according to the aggregate of dose-limiting toxicity criteria and adverse event (AE) data, and considering further pharmacokinetic and efficacy data of the derazantinib-paclitaxel-ramucirumab combination in patients with FGFR fusions, amplifications or mutations GAC.
Time Frame: From first dose and up to 18 months
Population: The Maximum Tolerated Dose (MTD)-determining population comprised all patients enrolled in Substudy 2 who meet the minimum criteria during the first 28-day treatment cycle (Cycle 1):
  * received at least one dose of derazantinib-paclitaxel-ramucirumab in combination and has experienced a DLT
  * or
  * received ≥ 80% of the derazantinib-paclitaxel-ramucirumab dose, respectively, in Cycle 1 and, had been observed for ≥ 28 days following the first dose, and had been evaluated for safety.
Measure: Number; unit: mg
Groups:
- Substudy 2 Combined: Derazantinib +Paclitaxel+ Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of either 200 mg or 300 mg once daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 2 Combined: Derazantinib +Paclitaxel+ Ramucirumab
Number analyzed (Participants) | 13
mg | 200

4. Secondary Outcome: ORR in Substudy 1 in Cohort 1.3
Description: ORR was defined by the percentage of patients with CR or PR by BICR according to RECIST Version 1.1.
Time Frame: From first dose and up to 9 months
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 13
Percentage of participants | 0.0 [0.0 to 20.6]

5. Secondary Outcome: Disease Control Rate (DCR) in Substudy 1: Cohort 1.1, 1.2 and 1.3 and Combined Cohorts
Description: Defined as the percentage of patients with confirmed CR, PR or stable disease (SD) by BICR per RECIST version 1.1.
Time Frame: From first dose and up to 18 months
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Substudy 1 Combined: Derazantinib 300 mg Once Daily or 200 mg Twice Daily: Derazantinib was administered orally at a dose of either 300 mg once daily or at a dose of 200 mg twice daily as monotherapy in Substudy 1.
Arm/Group | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily | Substudy 1 Combined: Derazantinib 300 mg Once Daily or 200 mg Twice Daily
Number analyzed (Participants) | 13 | 8 | 13 | 34
Percentage of participants | 30.8 [11.3 to 57.3] | 25.0 [4.6 to 60.0] | 15.4 [2.8 to 41.0] | 23.5 [12.3 to 38.5]

6. Secondary Outcome: PFS in Substudy 1 in Cohort 1.3
Description: PFS was calculated from patient enrollment to progressive disease (PD) date by BICR per RECIST version 1.1
Time Frame: From first dose and up to 9 months
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 13
months | 1.7 [1.0 to 1.9]

7. Secondary Outcome: Overall Survival (OS) in Substudy 1 in Cohort 1.3
Description: OS was measured from patient enrollment to time of death.
Time Frame: From first dose and up to 9 months
Population: The intent-to-treat (ITT) population comprised all patients enrolled and allocated to treatment, regardless of the administration of the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily: Derazantinib was administered orally at a dose of 200 mg twice daily as monotherapy in Substudy 1.
Arm/Group | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily
Number analyzed (Participants) | 13
months | 3.3 [2.2 to 3.7]

8. Secondary Outcome: OS in Substudy 2
Description: OS was measured from patient enrollment to time of death
Time Frame: From first dose and up to 15 months
Population: ITT population comprised all patients enrolled and allocated to treatment, regardless of the administration of the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Substudy 2: Derazantinib 300 mg Once Daily + Paclitaxel + Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of 300 mg once daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily + Paclitaxel + Ramucirumab
Number analyzed (Participants) | 6 | 7
months | 5.5 [2.7 to NA] — Not evaluable due to the low number of events. | NA [NA to NA] — Not evaluable due to the low number of events.

9. Secondary Outcome: ORR in Substudy 2
Description: ORR was defined by the percentage of patients with CR or PR by BICR per RECIST version 1.1.
Time Frame: From first dose and up to 15 months
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of 300 mg once daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab
Number analyzed (Participants) | 5 | 7
Percentage of participants | 40.0 [7.6 to 81.1] | 57.1 [22.5 to 87.1]

10. Secondary Outcome: DCR in Substudy 2
Description: Defined as the percentage of patients with confirmed CR, PR or SD by BICR per RECIST version 1.1.
Time Frame: From first dose and up to 15 months
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel + Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of 300 mg once daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel + Ramucirumab | Substudy 2 Combined: Derazantinib +Paclitaxel+ Ramucirumab
Number analyzed (Participants) | 5 | 7 | 12
Percentage of participants | 80.0 [34.3 to 99.0] | 71.4 [34.1 to 94.7] | 75.0 [47.3 to 92.8]

11. Secondary Outcome: DOR in Substudy 2 (Separate and Combined Cohorts)
Description: DOR was calculated from the first date of documented tumor response to disease progression by BICR per RECIST version 1.1 (or death if no documentation of PD is obtained).
Time Frame: From first dose and up to 15 months
Population: mITT population: all patients who received at least one dose of derazantinib and had at least one post-baseline imaging assessment in accordance with RECIST 1.1 or documented clinical progression or died from any cause on or after the first dose of study treatment and until safety follow-up visit (inclusive).
  Within the mITT, only patients with confirmed CR or PR have been considered for this endpoint (2 and 4 patients from the 200 mg and 300 mg arm, respectively)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of either 300 mg once daily or 200 mg twice daily in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2 Combined: Derazantinib +Paclitaxel+ Ramucirumab
Number analyzed (Participants) | 2 | 4 | 6
months | 9.2 [NA to NA] — Only a low number of patients with CR or PR (2 patients) and low number of related events (high number of censoring and time of censoring) could be considered for the evaluation. As such, some parameters are impossible to be estimated or to be evaluated by the statistical method used (Kaplan-Meier). | NA [3.3 to NA] — Only a low number of patients with CR or PR (4 patients) and low number of related events (high number of censoring and time of censoring) could be considered for the evaluation. As such, some parameters are impossible to be estimated or to be evaluated by the statistical method used (Kaplan-Meier). | 9.2 [3.3 to NA] — Only a low number of patients with CR or PR (2 and 4 patients from the 200 mg and 300 mg arm, respectively) and low number of related events (high number of censoring and time of censoring) could be considered for the evaluation. As such, some parameters are impossible to be estimated or to be evaluated by the statistical method used (Kaplan-Meier).

12. Secondary Outcome: PFS in Substudy 2
Description: PFS was calculated from patient enrollment to progressive disease (PD) date by BICR per RECIST version 1.1.
Time Frame: From first dose and up to 15 months
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab: Derazantinib-paclitaxel-ramucirumab combination: Derazantinib was administered orally at a dose of 300 mg in combination with paclitaxel and ramucirumab.
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab
Number analyzed (Participants) | 5 | 7
months | 11.1 [1.6 to NA] — Not evaluable due to the low number of events. | NA [1.7 to NA] — Not evaluable due to the low number of events.

13. Secondary Outcome: Number of Patients With at Least Grade 3 Treatment-emergent Adverse Events (TEAEs)
Description: Number of patients experiencing TEAE of Grade 3 and above according to Common Terminology Criteria for Adverse Events (CTCAE). CTCAE are a set of criteria for the standardized classification of TEAEs of drugs used in cancer therapy. It uses a range of grades from 1 to 5 describing increasing levels of severity of the TEAEs.
Time Frame: TEAEs defined as AEs which were assessed per patient from the patient's first dose and until 90 days after the last dose, which corresponded up to 19 months
Population: The Safety population comprises all patients who received at least one dose of study treatment (derazantinib, paclitaxel or ramucirumab).
Measure: Number; unit: Counts of participants
Arm/Group | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab
Number analyzed (Participants) | 13 | 8 | 13 | 6 | 7
Counts of participants
  Number of patients with only unrelated TEAEs of Grade 3 or above | 9 | 3 | 5 | 1 | 1
  Number of patients with related TEAEs of Grade 3 or above | 0 | 3 | 6 | 4 | 6
  Number of patients without TEAEs of Grade 3 or above | 4 | 2 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs which were assessed per patient from the patient's first dose and until 90 days after the last dose, which corresponded up to 19 months
Description: Treatment emergent adverse events (TEAEs) were defined as AEs that started or worsened in severity on or after the first dose of study treatment and until safety follow-up visit (inclusive).
Groups:
- Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab: Patients with FGFR fusions, amplifications or mutations were treated with 200 mg Derazantinib once daily in combination with Paclitaxel and Ramucirumab
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
- Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab: Patients with FGFR fusions, amplifications or mutations were treated with 300 mg Derazantinib once daily in combination with Paclitaxel and Ramucirumab
  Paclitaxel was administered intravenously at a dose of 80 mg/m² on days 1, 8, and 15 of a 28-day cycle in combination with ramucirumab.
  Ramucirumab was administered intravenously at a dose of 8 mg/kg every 2 weeks in combination with paclitaxel.
Arm/Group | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab
All-Cause Mortality (participants affected / at risk) | 10/13 | 6/8 | 10/13 | 4/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 7/13 | 4/8 | 10/13 | 4/6 | 3/7
Other Adverse Events (participants affected / at risk) | 12/13 | 8/8 | 13/13 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily (N=13) | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily (N=8) | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily (N=13) | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab (N=6) | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab (N=7)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 3 (3) | 2 (2) | 6 (6) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1: Cohort 1.1 Derazantinib 300 mg Once Daily (N=13) | Substudy 1: Cohort 1.2 Derazantinib 300 mg Once Daily (N=8) | Substudy 1: Cohort 1.3 Derazantinib 200 mg Twice Daily (N=13) | Substudy 2: Derazantinib 200 mg Once Daily +Paclitaxel+ Ramucirumab (N=6) | Substudy 2: Derazantinib 300 mg Once Daily +Paclitaxel+ Ramucirumab (N=7)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 6 (6) | 2 (2) | 5 (7)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 7 (9) | 3 (4) | 4 (7)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 5 (5) | 1 (1) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 2 (14)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 4 (4) | 3 (5) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Punctate keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 3 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (6) | 2 (2) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 6 (6) | 1 (1) | 1 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 0 (0) | 1 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 3 (4)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (3) | 5 (5) | 2 (2) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Penile haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT04604132/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT04604132/SAP_001.pdf